CLINICAL TRIAL: NCT00976560
Title: A Six Week Randomized, Double-blind, Multi-center, Placebo-controlled, Exploratory, Adaptive Design Study to Explore the Antidepressant Properties of the p38 MAP Kinase Inhibitor GW856553 Compared to Placebo in Adult Subjects With Major Depressive Disorder
Brief Title: Clinical Study to Test a New Drug to Treat Major Depression
Acronym: PKI113009
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113009
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Depressive Disorder, Major
Keywords: Lack of interest and energy; Psychomotor retardation; Cytokines; Major Depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Psychomotor Disorders | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GW856553 (Experimental): GW856553 7.5 mg BID
  Interventions: Drug: GW856553
- Placebo (Placebo Comparator): Matching Placebo BID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GW856553 — Wet Granulated, film coated white, 9mm round, biconvex, plain faced tablets, containing 7.5 mg of GW856553
  Arms: GW856553
Other: Placebo — Film coated white, 9mm round, biconvex, plain faced tablets obtained by direct compression.
  Arms: Placebo

SUMMARY:
In this randomized, double-blind, multi-centre, placebo controlled, exploratory, adaptive design study, the antidepressant and plasma cytokine lowering effects of the GW856553 will be investigated in adult subjects diagnosed with MDD. Subjects will receive oral doses of GW856553 or placebo for six weeks. Safety, tolerability, pharmacokinetics and pharmacodynamics, defined as biomarkers in blood and clinical symptoms, will be assessed.

The primary endpoint is the change from baseline associated with GW856553 versus placebo at Week 6 in the Bech (6-item HAMD-17) score. Interim analyses of the primary endpoint will be performed throughout the study to potentially adapt the study design by changing the randomization ratio and/ or reducing the total number of subjects to be randomized into the study. Exploratory analyses will be performed by associating changes in cytokine levels and selected clinical symptoms; PK/PD modelling will also be used to identify the most sensitive clinical and biological markers.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult subjects with primary diagnosis of moderate to severe MDD without psychotic features, for at least 4 weeks and one previous MDD episode
* Males or Females who agree to use protocol specified contraception if of child bearing potential
* BMI 18.5-35.0 kg/m2
* Normal liver function tests

Key Exclusion Criteria:

* History of liver disease or positive hepatitis B surface antigen or hepatitis C antibody in the last 3 months
* Elevated liver function tests on >2 ocassions in the last 7 months
* Significant medical illness, autoimmune disease or infectious disease
* Pregnant or nursing females
* Excessive and regular alcohol consumption
* History of substance abuse or dependence in past 6 months or positive urine drug screen
* Significant suicidal or homicidal risk
* Currently receiving chronic biological or pharmacologic anti-inflammatory therapy or is not euthyroid
* Psychoactive drugs within 1 week or 5 half lives of randomization visit
* Treatment resistant subjects

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2010-07-07 (Actual); Study Completion 2010-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (4):
  - GSK Investigational Site, Hoffman Estates, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Columbus, Ohio
- Bulgaria (4):
  - GSK Investigational Site, Pazardzhik
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
- GSK Investigational Site, Tartu, Estonia
- Germany (7):
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Westerstede, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Smolensk

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 25 Sep 2009 to 7 July 2010. The study was conducted at 21 centers in 5 countries (Bulgaria [4], Estonia [1], Germany [7], Russia [5], United States [4]).
Pre-assignment Details: A total of 128 participants of both the gender, with major depressive disorder (MDD), having at least one previous major depressive episode in history and currently undergoing a recurrence, of age group 18 to 60, were enrolled globally. A total of 231 participants were screened of which 103 were screen-failures.
Groups:
- Placebo: Eligible participants received matching placebo, orally, twice daily with food at morning and evening with the interval of 12 hours for 6 weeks.
- GW856553 7.5 mg BID: Eligible participants received GW856553 7.5 mg, orally, twice daily with food at morning and evening with the interval of 12 hours for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | GW856553 7.5 mg BID
Started | 64 | 64
Completed | 50 | 51
Not Completed | 14 | 13
Not completed — Adverse Event | 5 | 5
Not completed — Lack of Efficacy | 3 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GW856553 7.5 mg BID | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Customized [Count of Participants; unit: Participants]
  18 to 60 years | 64 | 64 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 76
  Male | 27 | 25 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 60 | 63 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization (Week 0) Associated With GW856553 Versus Placebo at Week 6 in the Bech (6-item HAMD-17 [Hamilton Depression Rating Scale]) Score.
Description: HAMD-17 has 17 questions. The HAMD-17 Total Score was calculated by summing the individual response scores over the 17 individual components of the interview. The highest possible score was 52, which represented the most severe measure of depression; the lowest possible score was 0, which represented an absence of depression. There were 9 five point questions and 8 three point questions. The responses to the individual questions had values of 0-2 (three points response) or 0-4 (five points response). The BECH scale was extracted from the HAMD-17 and comprises of 6 items out of which 5 are 5 point questions and 1 is 3 point question. The Bech Total Score was calculated by summing the individual response scores and ranged from 0 to 22, with higher scores indicating more severe depression. Week 0 values were considered as Baseline.The change from randomization was analysed using suitable Bayesian mixed-effects model repeated measures (BMMRM) assuming missing at random (MAR).
Time Frame: At Week 6
Population: Intent-to-Treat (ITT) - It comprised of all randomised participants who received at least one dose of study medication and had at least one post-dose efficacy assessment.
  Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 50 | 51
Scores on scale | -6.5 (3.62) | -5.6 (3.74)
Statistical Analysis 1: Comparison: Placebo vs GW856553 7.5 mg BID; Test type: Superiority or Other; BMMRM; Bayesian Mixed Effects Model Repeated Measures (BMMRM); Mean Difference (Net) = -0.60, 95% CI 2-sided [-2.54 to 1.35], Standard Deviation 0.990 — Prior distribution of N(-4.1, 6.4009) incorporated into the posterior for the treatment difference at Week 6. The presented Confidence Interval is Highest Probability Density (HPD); Posterior probability of the treatment difference being greater than 1.6 points in favor of GW856553 7.5mg BID as compared to placebo at Week 6 is 15.46 and for 0 is 72.98 and for 2 is 7.87

2. Secondary Outcome: Number of Participants With Adverse Events
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A Serious Adverse Event (SAE) is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. The AEs row include participants with SAEs.
Time Frame: 6 Weeks
Population: All Subjects Population - It comprised of all participants who receive at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 64 | 64
Participants
  AEs | 28 | 26
  SAEs | 1 | 1

3. Secondary Outcome: Number of Participants With Suicidality as Assessed by the Columbia Suicidality Severity Rating Scale Score
Description: Suicidility was defined as participants with major depressive disorder who experienced worsening of their depression and/or the emergence of suicidal ideation and behavior. Number of partcipants who experienced suicidality were reported. On the Suicidal Ideation scale of the Columbia Suicide-Severity Rating Scale (C-SSRS) participants were scored as "non-suicidal" (00), "wish to be dead" (01), "non-specific active suicidal thoughts" (02), "active suicidal ideation with associated thoughts of methods without intent" (03), "active suicidal ideation with some intent to act on suicidal thoughts without clear plan" (04) and "active suicidal ideation with plan and intent" (05), based on the most severe score (5 being the most severe).Suicidal ideation of type 4 or 5 in the C-SSRS was categorized as suicidility here.
Time Frame: Upto Week 6
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 64 | 64
Participants
  Week 1, Non-suicidal: number analyzed (Participants) | 55 | 57
  Week 1, Non-suicidal | 55 | 57
  Week 2, Non-suicidal: number analyzed (Participants) | 54 | 55
  Week 2, Non-suicidal | 54 | 55
  Week 3, Non-suicidal: number analyzed (Participants) | 49 | 54
  Week 3, Non-suicidal | 49 | 54
  Week 4, Non-suicidal: number analyzed (Participants) | 50 | 54
  Week 4, Non-suicidal | 50 | 54
  Week 5, Non-suicidal: number analyzed (Participants) | 49 | 50
  Week 5, Non-suicidal | 49 | 50
  Week 6, Non-suicidal: number analyzed (Participants) | 50 | 49
  Week 6, Non-suicidal | 50 | 49

4. Secondary Outcome: Number of Participants With Abnormal Haematology and Clinical Chemistry Values
Description: Samples for haematology and clinical chemistry were collected on Weeks 1, 5 and 6. The analyzed haematological parameters were platelet count, red blood cells count, white blood cells count, reticulocyte count, hemoglobin and hematocrit. The analyzed clinical chemistry parameters were urea, creatinine, glucose (fasting), sodium, lactate dehydrogenase (LDH), potassium, chloride, calcium, triglycerides, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), alkaline phosphatase, creatine kinase (CK), total and direct bilirubin, albumin, total protein and total cholesterol. Number of participants with any abnormal haematological or clinical chemistry parametrs are summarized here.
Time Frame: Upto Week 6
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 64 | 64
Participants
  Glucose High, Week 6: number analyzed (Participants) | 44 | 46
  Glucose High, Week 6 | 1 | 0
  Total Bilirubin High, Week 4: number analyzed (Participants) | 45 | 51
  Total Bilirubin High, Week 4 | 1 | 0

5. Secondary Outcome: Number of Participants With Abnormal Vital Signs (Blood Pressure, Heart Rate)
Description: Vital signs including systolic and diastolic blood pressure and heart rate were taken from day 1 upto follow-up visit. Number of participants with abnormal systolic blood pressure, diastolic blood pressure and heart rate values were summarized.
Time Frame: Up to follow-up Visit (Day 53)
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 64 | 64
Participants
  Low Diastolic blood pressure, Week 4: number analyzed (Participants) | 53 | 56
  Low Diastolic blood pressure, Week 4 | 1 | 0
  High Systolic blood pressure, Week 2: number analyzed (Participants) | 59 | 60
  High Systolic blood pressure, Week 2 | 1 | 0

6. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: ECG was obtained at Week 2 and Week 6. ECG was recorded using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and Corrected QT (QTc) intervals (Bazett's correction was applied to QTc measurements). Number of participants with abnormal ECG readings are summarized.
Time Frame: Up to follow-up Visit (Day 53)
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 64 | 64
Participants | 0 | 0

7. Secondary Outcome: Changes From Randomization (Week 0)in IL-6 and TNF-alpha Associated With GW856553 Versus Placebo at Week 1 and Week 6 in the Morning Plasma Levels
Description: Interlukin-6 (IL-6) and Tumor Necrosis Factor-Alpha (TNF-alpha) from the participants with Major Depressive Disorder (MDD) were evaluated and analyzed using suitable mixed-effects model repeated measures (MMRM). Exploratory analysis on plasma levels of IL-6 and TNF-alpha were performed. Week 0 values were considered as Baseline.The change from Baseline was calculated by subtracting the baseline values from the individual post-randomisation values.
Time Frame: Upto Week 6
Population: Intent-to-Treat (ITT) Population - It consists of all randomised subjects who receive at least one dose of study medication and had at least one post-dose efficacy assessment.
  Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: picogram/mililitre (pg/mL)
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 62 | 63
picogram/mililitre (pg/mL)
  IL-6, Week 1, Predose: number analyzed (Participants) | 58 | 62
  IL-6, Week 1, Predose | -1.06 (8.04) | -0.27 (4.36)
  IL-6, Week 1, 3 hours (hrs): number analyzed (Participants) | 61 | 63
  IL-6, Week 1, 3 hours (hrs) | -1.86 (9.72) | -1.57 (4.30)
  IL-6, Week 6, Predose: number analyzed (Participants) | 50 | 51
  IL-6, Week 6, Predose | -0.67 (11.29) | -0.96 (5.68)
  IL-6, Week 6, 3 hrs: number analyzed (Participants) | 50 | 51
  IL-6, Week 6, 3 hrs | -0.11 (8.93) | -0.98 (9.36)
  IL-6, Early Withdrawal: number analyzed (Participants) | 9 | 11
  IL-6, Early Withdrawal | -7.44 (15.54) | 0.35 (4.52)
  TNF-alpha, Week 1, Predose: number analyzed (Participants) | 56 | 60
  TNF-alpha, Week 1, Predose | 1.04 (9.65) | -0.26 (1.43)
  TNF-alpha, Week 1, 3 hrs: number analyzed (Participants) | 59 | 60
  TNF-alpha, Week 1, 3 hrs | 1.41 (12.61) | -0.65 (1.61)
  TNF-alpha, Week 6, Predose: number analyzed (Participants) | 48 | 49
  TNF-alpha, Week 6, Predose | 3.80 (28.78) | -0.10 (1.57)
  TNF-alpha, Week 6, 3 hrs: number analyzed (Participants) | 49 | 49
  TNF-alpha, Week 6, 3 hrs | 4.11 (29.20) | -0.63 (1.49)
  TNF-alpha, Eary Withdrawal: number analyzed (Participants) | 9 | 11
  TNF-alpha, Eary Withdrawal | 0.31 (0.96) | -1.07 (2.24)

8. Secondary Outcome: Change From Randomisation Bech Total Score: Bech Score
Description: HAMD-17 has 17 questions. The BECH scale was extracted from the HAMD-17 and comprises of 6 items out of which 5 are 5 point questions and 1 is 3 point question. The Bech scale was extracted from the HAMD-17 and comprised of 6 items out of which 5 were 5 point questions and 1 was 3 point question. The Bech Total Score was calculated by summing the individual response scores and ranged from 0 to 22, with higher scores indicating more severe depression. Due to the small number of items, missing data was not imputed for the Bech Total Score. If any of the 6 items were missing, the total score was not calculated at that visit. The change from randomization was analysed using suitable Bayesian Mixed-Effects Models for Repeated Measures (BMMRM) assuming missing at random MAR.
Time Frame: Up to Follow-up visit (Day 53)
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 62 | 63
Scores on scale
  Week 1 | -1.2 (2.14) | -1.6 (2.47)
  Week 2: number analyzed (Participants) | 59 | 60
  Week 2 | -2.5 (2.73) | -2.2 (2.91)
  Week 3: number analyzed (Participants) | 54 | 58
  Week 3 | -3.9 (3.20) | -3.4 (3.07)
  Week 4: number analyzed (Participants) | 53 | 57
  Week 4 | -5.1 (2.97) | -4.1 (3.43)
  Week 5: number analyzed (Participants) | 52 | 54
  Week 5 | -6.2 (3.49) | -5.0 (3.60)
  Week 6: number analyzed (Participants) | 50 | 51
  Week 6 | -6.5 (3.62) | -5.6 (3.74)
  Follow Up: number analyzed (Participants) | 60 | 61
  Follow Up | -5.6 (3.58) | -5.2 (4.12)
  Early Withdrawal: number analyzed (Participants) | 4 | 6
  Early Withdrawal | 0.3 (1.26) | -2.0 (4.00)

9. Secondary Outcome: Mean HAMD-17 Total Score
Description: HAMD-17 is Hamilton Depression Rating Scale which has 17 questions. The HAMD-17 Total Score was calculated by summing the individual response scores over the 17 individual components of the interview. The highest possible score was 52, which represented the most severe measure of depression; the lowest possible score was 0, which represented an absence of depression. If not more than 1 response was missing, the total score was caculated as Observed Total Score * [1 + (Sum of the Maximum Score of the missing values/Sum of the Maximum Score of the non -missing values)]. There were 9 five point questions and 8 three point questions. The responses to the individual questions can have values of 0-2 (three points response) or 0-4 (five points response).
Time Frame: Up to Follow-up visit (Day 53)
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 62 | 63
Scores on Scale
  Week 1 | 21.7 (4.88) | 21.2 (4.78)
  Week 2: number analyzed (Participants) | 59 | 60
  Week 2 | 18.9 (5.59) | 19.7 (5.36)
  Week 3: number analyzed (Participants) | 54 | 58
  Week 3 | 16.5 (6.76) | 17.8 (5.57)
  Week 4: number analyzed (Participants) | 53 | 57
  Week 4 | 14.1 (6.10) | 16.6 (5.39)
  Week 5: number analyzed (Participants) | 52 | 54
  Week 5 | 12.6 (7.43) | 14.8 (6.14)
  Week 6: number analyzed (Participants) | 50 | 51
  Week 6 | 11.7 (7.05) | 13.8 (6.50)
  Follow up: number analyzed (Participants) | 60 | 61
  Follow up | 13.4 (7.34) | 14.4 (7.41)
  Early Withdrawal: number analyzed (Participants) | 4 | 6
  Early Withdrawal | 27.8 (5.74) | 23.5 (4.18)

10. Secondary Outcome: Mean Inventory of Depressive Symptomatology Clinician (IDS-C) Total Score
Description: The 30 item IDS is available in two versions IDS-C and Inventory of Depressive Symptomatology self-rated (IDS-SR). To calculate the total score of IDS, 28 out of the 30 items were scored. Either weight loss or weight gain, appetite loss or appetite gain is scored because only one member of each pair is applicable to any given respondent. The standard total score is obtained by summing the ratings of 28 of the 30 items. Each of the 28 items is scored on a 0 to 3 scale (0 - the absence of pathology; 3 - severe pathology). The total scores range from 0 to 84. If more than one response was missing then the score was calculated using the formula Observed Total Score*[1+(Sum of the Maximum Score of the missing values/Sum of the Maximum Score of the non -missing values)].
Time Frame: Up to Follow-up visit (Day 53)
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 62 | 63
Scores on Scale
  Week1 | 39.7 (8.7) | 39.2 (8.5)
  Week 2: number analyzed (Participants) | 59 | 60
  Week 2 | 35.2 (9.8) | 35.9 (9.1)
  Week 3: number analyzed (Participants) | 54 | 58
  Week 3 | 30.9 (11.8) | 32.4 (9.3)
  Week 4: number analyzed (Participants) | 53 | 57
  Week 4 | 26.9 (10.7) | 30.9 (9.8)
  Week 5: number analyzed (Participants) | 52 | 54
  Week 5 | 23.4 (13.5) | 27.1 (11.3)
  Week 6: number analyzed (Participants) | 50 | 51
  Week 6 | 22.0 (12.8) | 25.8 (12.1)
  Follow-up: number analyzed (Participants) | 60 | 61
  Follow-up | 25.3 (13.6) | 26.6 (12.8)
  Early Withdrawal: number analyzed (Participants) | 4 | 6
  Early Withdrawal | 47.0 (13.5) | 41.8 (7.0)

11. Secondary Outcome: Mean IDS-SR Total Score
Description: The 30 item IDS is available in two versions IDS-SR and IDS-C. To calculate the total score of IDS, 28 out of the 30 items were scored. Either weight loss or weight gain, appetite loss or appetite gain is scored because only one member of each pair is applicable to any given respondent. The standard total score is obtained by summing the ratings of 28 of the 30 items. Each of the 28 items is scored on a 0 to 3 scale (0 - the absence of pathology; 3 - severe pathology). The total scores range from 0 to 84. If more than one response was missing then the score was calculated using the formula Observed Total Score*[1+(Sum of the Maximum Score of the missing values/Sum of the Maximum Score of the non -missing values)].
Time Frame: Up to Week 6
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 62 | 63
Scores on Scale
  Week 2: number analyzed (Participants) | 61 | 61
  Week 2 | 34.7 (11.02) | 38.1 (10.79)
  Week 4: number analyzed (Participants) | 56 | 58
  Week 4 | 29.2 (11.84) | 32.8 (12.15)
  Week 6: number analyzed (Participants) | 51 | 53
  Week 6 | 24.7 (14.98) | 27.5 (13.28)
  Early Termination: number analyzed (Participants) | 4 | 6
  Early Termination | 48.8 (14.13) | 47.0 (10.64)

12. Secondary Outcome: Mean Quick Inventory of Depressive Symptomatology Self Report-16 Item (QIDS-SR16) Total Score Derived From the IDS-SR (Only at Weeks 0, 2, 4 and 6)
Description: QIDS-SR assesses symptoms severity of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criterion for major depressive disorder. It contains 16 separate items (corresponding to 16 items of the much longer IDS-SR), defining 9 DSM-IV symptom criterion domains. A total score was obtained by summing scores on each domain. The QIDS-SR total score was calculated by summing over the domain scores. The highest possible score was 27, which represented the most severe measure of depression; the lowest possible score was 0, which represented an absence of depression. Due to the small number of items, missing data was not imputed for the QIDS-SR total score.
Time Frame: Weeks 0, 2, 4 and 6
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 62 | 63
Scores on Scale
  Week 0 | 18.0 (2.79) | 17.8 (2.66)
  Week 2: number analyzed (Participants) | 61 | 61
  Week 2 | 13.0 (4.22) | 14.1 (3.99)
  Week 4: number analyzed (Participants) | 56 | 58
  Week 4 | 10.6 (4.69) | 11.8 (4.46)
  Week 6: number analyzed (Participants) | 51 | 53
  Week 6 | 9.3 (5.81) | 10.0 (4.75)

13. Secondary Outcome: Percentage of IDS-C Responders (Participants With a Reduction in Total Score of ≥50% From Randomization at Week 6/Study Exit).
Description: The 30 item IDS is available in two versions IDS-C and IDS-SR. To calculate the total score of IDS, 28 out of the 30 items were scored. Either item 11 or 12 (and 13 or 14) were scored. If 11 and 12 (or 13 and 14) both are scored then the item with the highest score was considered. The total score of the 28 items ranged between 0-84. A responder is a participant who has a ≥50% reduction from randomisation in the total score for IDS-C. The total score was calculated for each participant at each timepoint and the percentage change from randomisation was then calculated as ([Total score at post randomisation visit - Total score at randomisation visit]/ Total score at randomisation visit) * 100%. Responders were those with values of ≤ -50%. The change from randomization was analysed using suitable Bayesian mixed-effects model repeated measures (BMMRM) assuming missing at random (MAR).
Time Frame: Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 50 | 51
Percentage of Participants | 50 | 41

14. Secondary Outcome: Percentage of IDS-C Remitters (Participants Whose Total Score Was ≤ 15 at Week 6/Study Exit).
Description: The 30 item IDS is available in two versions IDS-C and IDS-SR. To calculate the total score of IDS, 28 out of the 30 items were scored. Either item 11 or 12 (and 13 or 14) were scored. If 11 and 12 (or 13 and 14) both are scored then the item with the highest score was considered. The total score of the 28 items ranged between 0-84. IDS-C total score was calculated for each participant at each timepoint and those participants with non-missing values for IDS-C total scores were categorised as having an IDS-C for the respective endpoint of ≤ 15 or > 15. Participants whose total score was ≤ 15 were included here.
Time Frame: Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 50 | 51
Percentage of participants | 38 | 18

15. Secondary Outcome: Percentage of IDS-SR Responders (Participants With a Reduction in Total Score of ≥ 50% From Randomization at Week 6/Study Exit).
Description: The 30 item IDS is available in two versions IDS-C and IDS-SR. To calculate the total score of IDS, 28 out of the 30 items were scored. Either item 11 or 12 (and 13 or 14) were scored. If 11 and 12 (or 13 and 14) both are scored then the item with the highest score was considered. The total score of the 28 items ranged between 0-84. A responder is a participant who has a ≥50% reduction from randomisation in the total score for IDS-SR. The total score was calculated for each participant at each timepoint and the percentage change from randomisation was then calculated as ([Total score at post randomisation visit - Total score at randomisation visit]/ Total score at randomisation visit) * 100%. Responders were those with values of ≤ -50%. The change from randomization was analysed using suitable BMMRM assuming missing at random.
Time Frame: Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 51 | 53
Participants | 49 | 47

16. Secondary Outcome: Percentage of IDS-SR Remitters (Participants Whose Total Score Was ≤ 15 at Week 6/Study Exit).
Description: The 30 item IDS is available in two versions IDS-C and IDS-SR. To calculate the total score of IDS, 28 out of the 30 items were scored. Either item 11 or 12 (and 13 or 14) were scored. If 11 and 12 (or 13 and 14) both are scored then the item with the highest score was considered. The total score of the 28 items ranged between 0-84. IDS-SR total score was calculated for each participant at each timepoint and those participants with non-missing values for IDS-SR total scores were categorised as having an IDS-C for the respective endpoint of ≤ 15 or > 15. Participants whose total score was ≤ 15 were included here.
Time Frame: Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 51 | 53
Percentage of participants | 37 | 19

17. Secondary Outcome: Percentage of QIDS-SR16 Responders (Participants With a Reduction in Total Score of ≥ 50% From Randomization at Week 6/Study Exit).
Description: QIDS-SR assesses symptoms severity of DSM-IV diagnostic criterion for major depressive disorder. It contains 16 separate items (corresponding to 16 items of the much longer IDS-SR), defining 9 DSM-IV symptom criterion domains. A total score was obtained by summing scores on each domain.The highest possible score was 27, which represented the most severe measure of depression; the lowest possible score was 0, which represented an absence of depression. Due to the small number of items, missing data was not imputed for the QIDS-SR total score. A responder is a participant who has a ≥50% reduction from randomisation in the total score for that given endpoint. The total score was calculated for each participant at each timepoint and the percentage change from randomisation was then calculated as ([Total score at post randomisation visit - Total score at randomisation visit]/ Total score at randomisation visit) * 100%. Responders were those with values of ≤ -50%.
Time Frame: Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 51 | 53
Percentage of Participants | 55 | 45

18. Secondary Outcome: Percentage of QIDS-SR16 Remitters (Subjects Whose Total Score Was ≤ 5 at Week 6/Study Exit).
Description: QIDS-SR assesses symptoms severity of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criterion for major depressive disorder. It contains 16 separate items (corresponding to 16 items of the much longer IDS-SR), defining 9 DSM-IV symptom criterion domains. A total score was obtained by summing scores on each domain. The QIDS-SR total score was calculated by summing over the domain scores. The highest possible score was 27, which represented the most severe measure of depression; the lowest possible score was 0, which represented an absence of depression. Due to the small number of items, missing data was not imputed for the QIDS-SR total score. The QIDS total score was calculated for each subject at each timepoint and those subjects with no missing value for QIDS total score was categorised as having a QIDS total score of ≤ 5 or > 5. Participants whose total score was ≤ 5 were included here.
Time Frame: Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 51 | 53
Percentage of participants | 31 | 13

19. Secondary Outcome: Percentage of Bech Responders (Participants With a Reduction in Total Score of ≥ 50% From Randomization at Week 6/Study Exit).
Description: The Bech scale was extracted from the HAMD-17 and comprised of 6 items out of which 5 were 5 point questions and 1 was 3 point question. The Bech Total Score was calculated by summing the individual response scores. Due to the small number of items, missing data was not imputed for the Bech Total Score. If any of the 6 items were missing, the total score was not calculated at that visit. A responder is a participant who has a ≥50% reduction from randomisation in the total score for that given endpoint. The total score was calculated for each participant at each timepoint and the percentage change from randomisation was then calculated as ([Total score at post randomisation visit - Total score at randomisation visit]/ Total score at randomisation visit) * 100%. Responders were those with values of ≤ -50%. The change from randomization was analysed using suitable BMMRM assuming missing at random.
Time Frame: Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 51 | 50
Percentage of participants | 62 | 49

20. Secondary Outcome: Percentage of Bech Remitters (Participants Whose Total Score Was ≤ 4 at Week 6/Study Exit).
Description: The Bech scale was extracted from the HAMD-17 and comprised of 6 items out of which 5 were 5 point questions and 1 was 3 point question. The Bech Total Score was calculated by summing the individual response scores. Due to the small number of items, missing data was not imputed for the Bech Total Score. If any of the 6 items were missing, the total score was not calculated at that visit. The change from randomization was analysed using suitable BMMRM assuming missing at random MAR. The BECH total score was calculated for each subject at each timepoint and those perticipants with no missing value for BECH total score were categorised as having a BECH total score of ≤ 4 or > 4.
Time Frame: Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 51 | 50
Percentage of participants | 38 | 20

21. Secondary Outcome: Percentage of Participants With a Clinicians Global Impression of Improvement (CGI-I) Score of 1 ("Very Much Improved") or 2 ("Much Improved") at Weeks 1, 2, 3, 4, 5 and 6.
Description: The number of participantts with a CGI-I score of either 1 ("very much improved") or 2 (much improved") were grouped together for each timepoint. Participants with no missing CGI-I scores were categorised as having a CGI-I score of ≤ 2 or > 2.
Time Frame: Weeks 1, 2, 3, 4, 5 and 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 62 | 63
Percentage of participants
  Week 1: number analyzed (Participants) | 61 | 63
  Week 1 | 10 | 8
  Week 2: number analyzed (Participants) | 58 | 59
  Week 2 | 28 | 14
  Week 3: number analyzed (Participants) | 51 | 57
  Week 3 | 41 | 39
  Week 4: number analyzed (Participants) | 53 | 56
  Week 4 | 53 | 36
  Week 5: number analyzed (Participants) | 51 | 52
  Week 5 | 61 | 54
  Week 6: number analyzed (Participants) | 50 | 51
  Week 6 | 68 | 59

22. Secondary Outcome: Assessment of Clinical Global Impression-Severity of Illness (CGI-S) up to 6 Weeks
Description: CGI-S assesses the severity of the participant's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill). The number of participants with a CGI-I score of either 1 ("very much improved") or 2 (much improved") were grouped together for each timepoint. Participants with no missing CGI-S scores were categorised as having a CGI-S score of ≤ 2 or > 2. The total score was calculated for each participant at each timepoint and percentage was calculated.
Time Frame: Upto Week 6
Population: ITT Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW856553 7.5 mg BID
Number analyzed (Participants) | 62 | 63
Percentage of participants
  Week 1, Normal: number analyzed (Participants) | 61 | 63
  Week 1, Normal | 0 | 1.59
  Week 2, Normal: number analyzed (Participants) | 58 | 59
  Week 2, Normal | 0 | 1.69
  Week 3, Normal: number analyzed (Participants) | 51 | 57
  Week 3, Normal | 1.96 | 3.51
  Week 4, Normal: number analyzed (Participants) | 53 | 56
  Week 4, Normal | 0 | 1.79
  Week 5, Normal: number analyzed (Participants) | 51 | 52
  Week 5, Normal | 13.73 | 3.85
  Week 6, Normal: number analyzed (Participants) | 50 | 51
  Week 6, Normal | 12.00 | 3.92
  Week 1, Borderline Mentally ill: number analyzed (Participants) | 61 | 63
  Week 1, Borderline Mentally ill | 0 | 1.59
  Week 2, Borderline Mentally ill: number analyzed (Participants) | 58 | 59
  Week 2, Borderline Mentally ill | 3.45 | 3.39
  Week 3, Borderline Mentally ill: number analyzed (Participants) | 51 | 57
  Week 3, Borderline Mentally ill | 9.80 | 1.75
  Week 4, Borderline Mentally ill: number analyzed (Participants) | 53 | 56
  Week 4, Borderline Mentally ill | 16.98 | 7.14
  Week 5, Borderline Mentally ill: number analyzed (Participants) | 51 | 52
  Week 5, Borderline Mentally ill | 17.65 | 17.31
  Week 6, Borderline Mentally ill: number analyzed (Participants) | 50 | 51
  Week 6, Borderline Mentally ill | 20.00 | 23.53
  Week 1, Mildly ill: number analyzed (Participants) | 61 | 63
  Week 1, Mildly ill | 9.84 | 3.17
  Week 2, Mildly ill: number analyzed (Participants) | 58 | 59
  Week 2, Mildly ill | 18.97 | 6.78
  Week 3, Mildly ill: number analyzed (Participants) | 51 | 57
  Week 3, Mildly ill | 29.41 | 24.56
  Week 4, Mildly ill: number analyzed (Participants) | 53 | 56
  Week 4, Mildly ill | 41.51 | 26.79
  Week 5, Mildly ill: number analyzed (Participants) | 51 | 52
  Week 5, Mildly ill | 33.33 | 28.85
  Week 6, Mildly ill: number analyzed (Participants) | 50 | 51
  Week 6, Mildly ill | 34.00 | 29.41
  Week 1, Moderately ill: number analyzed (Participants) | 61 | 63
  Week 1, Moderately ill | 40.98 | 46.03
  Week 2, Moderately ill: number analyzed (Participants) | 58 | 59
  Week 2, Moderately ill | 46.55 | 50.85
  Week 3, Moderately ill: number analyzed (Participants) | 51 | 57
  Week 3, Moderately ill | 29.41 | 40.35
  Week 4, Moderately ill: number analyzed (Participants) | 53 | 56
  Week 4, Moderately ill | 22.64 | 39.29
  Week 5, Moderately ill: number analyzed (Participants) | 51 | 52
  Week 5, Moderately ill | 17.65 | 25.00
  Week 6, Moderately ill: number analyzed (Participants) | 50 | 51
  Week 6, Moderately ill | 20.00 | 19.61
  Week 1, Markedly ill: number analyzed (Participants) | 61 | 63
  Week 1, Markedly ill | 36.07 | 38.10
  Week 2, Markedly ill: number analyzed (Participants) | 58 | 59
  Week 2, Markedly ill | 20.69 | 30.51
  Week 3, Markedly ill: number analyzed (Participants) | 51 | 57
  Week 3, Markedly ill | 21.57 | 22.81
  Week 4, Markedly ill: number analyzed (Participants) | 53 | 56
  Week 4, Markedly ill | 16.98 | 19.64
  Week 5, Markedly ill: number analyzed (Participants) | 51 | 52
  Week 5, Markedly ill | 15.69 | 23.08
  Week 6, Markedly ill: number analyzed (Participants) | 50 | 51
  Week 6, Markedly ill | 10.00 | 21.57
  Week 1, Severely ill: number analyzed (Participants) | 61 | 63
  Week 1, Severely ill | 13.11 | 9.52
  Week 2, Severely ill: number analyzed (Participants) | 58 | 59
  Week 2, Severely ill | 10.34 | 6.78
  Week 3, Severely ill: number analyzed (Participants) | 51 | 57
  Week 3, Severely ill | 7.84 | 7.02
  Week 4, Severely ill: number analyzed (Participants) | 53 | 56
  Week 4, Severely ill | 1.89 | 5.36
  Week 5, Severely ill: number analyzed (Participants) | 51 | 52
  Week 5, Severely ill | 1.96 | 1.92
  Week 6, Severely ill: number analyzed (Participants) | 50 | 51
  Week 6, Severely ill | 4.00 | 1.96

ADVERSE EVENTS:
Time Frame: Up to Follow-up visit (Day 53).
Description: All SAEs and Non-SAEs were reported in All Subjects Population
Arm/Group | Placebo | GW856553 7.5 mg BID
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/64 | 1/64
Other Adverse Events (participants affected / at risk) | 18/64 | 16/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | GW856553 7.5 mg BID (N=64)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | GW856553 7.5 mg BID (N=64)
Headache (Nervous system disorders) | 9 | 12
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Anxiety (Psychiatric disorders) | 2 | 4
Fatigue (General disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.